CLINICAL TRIAL: NCT06030778
Title: HEALTHCARE STUDENTS' ATTITUDES TOWARDS PATIENTS WITH CHRONIC PAIN: VALIDITY AND RELIABILITY STUDY
Brief Title: HEALTHCARE STUDENTS' ATTITUDES TOWARDS PATIENTS WITH CHRONIC PAIN
Acronym: quantitative
Status: Completed | Type: Observational
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Nefise Cevriye SUCU ÇAKMAK, Dr., Çankırı Karatekin University
Other Study IDs: Nefise C. SUCU ÇAKMAK
Record Dates: First submitted 2023-09-03; First posted 2023-09-11 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Attitude to the Patient With Chronic Pain; Attitude of Health Care Students
Keywords: Nursing students; Healthcare students; Chronic pain; Attitude; Validity and reliability study
MeSH Terms: conditions — Chronic Pain; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention group: The descriptive characteristics form and the attitude scale of healthcare professionals towards their patients with chronic pain were administered to 205 students from the departments of medicine, physical therapy and rehabilitation, and nursing who agreed to participate in the study. The attitude scale of the health professionals towards their chronic pain patients was applied to 29 randomly selected students among these 205 students 15 days later.

SUMMARY:
Researchers studied the attitude towards patients with chronic pain, it is a very important issue for the literature. The prevalence of chronic pain is very high in the world, however, patients with chronic pain state at every opportunity that patients are not sufficiently understood and stigmatized by healthcare professionals. In this article, researchers studied the validity and reliability of the scale of the attitude of healthcare professionals towards their patients with chronic pain in students studying in the field of health (medicine, physical therapy and rehabilitation, nursing). Researchers found that the Healthcare Professionals' Attitudes towards Patients with Chronic Pain Scale was valid and reliable in healthcare students. Thanks to this scale, students' attitudes towards patients with chronic pain will be measured, and an idea will be gained about the student's deficiency.

ELIGIBILITY:
Inclusion Criteria:

Medicine, nursing, and physical therapy and rehabilitation students in their final year, With internet access, Who want to participate in the study.

Exclusion Criteria:

Medicine, nursing, and physical therapy and rehabilitation 1st, 2nd, and 3rd year undergraduate students Not wanting to participate in the research

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The final year students in the three healthcare departments of a university, namely medicine, nursing, and physical therapy and rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Healthcare Professionals' Attitudes towards Patients with Chronic Pain Scale's data | 1-29 january 2022
  reliability and validity findings

SECONDARY OUTCOMES:
Healthcare Professionals' Attitudes towards Patients with Chronic Pain Scale's remeasurement data | 1-15 february 2022
  test-retest findings

CONTACTS AND LOCATIONS:
Locations (1):
- Nefise Cevriye SUCU ÇAKMAK, Çankırı, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: for 5 years
Access Criteria: The data set can be shared as long as the author is requested via email.